CLINICAL TRIAL: NCT03704870
Title: A Randomized Controlled Feasibility Study Looking at Differences in Hospital Stay Variables Following Omission of Daily Routine Chest Radiographs After Pulmonary Resection.
Brief Title: Outcomes Following Omission of Daily Routine Chest Radiographs Following Pulmonary Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-5398
Record Dates: First submitted 2018-02-28; First posted 2018-10-15 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer; Lung Diseases; Lung Cancer, Nonsmall Cell; Surgery; Lung Adenocarcinoma
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Chest Xray (standard) (Active Comparator)
  Interventions: Diagnostic Test: Chest Xray
- Chest Xray post chest tube removal only (Experimental)
  Interventions: Diagnostic Test: No daily chest xray

INTERVENTIONS:
Diagnostic Test: Chest Xray — Daily chest xray
  Arms: Daily Chest Xray (standard)
Diagnostic Test: No daily chest xray — Chest xray will be done post chest tube removal only
  Arms: Chest Xray post chest tube removal only

SUMMARY:
Currently, it is the standard of care practice to perform daily routine CXR when a chest tube is in situ following pulmonary resection. However, previous research as well as experience of thoracic surgeons suggested this kind of management has poor diagnostic and therapeutic value. Eliminating daily routine CXR for adult patients having undergone pulmonary surgery might decrease the frequency of radiation exposure and hospitalization costs per patient without increasing reintervention rates, length of hospital stays, readmission rates or any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females who plan to receive VATS pulmonary resections confined to lobectomies, segmentectomies and wedge resections.
* Willingness to adhere to randomized treatment.
* Ability to answer self- and interviewer- administered questions in English
* Understand and sign a written informed consent form in English

Exclusion Criteria:

* Previous thoracic surgery history in the same side.
* Exploration, biopsy, lung volume reduction surgeries (LVRS), bilobectomies, sleeve resections or pneumonectomies performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of total chest xrays performed per subject | 30 days
  number of scheduled and additional chest xrays, and how does this correlate with post operative safety

CONTACTS AND LOCATIONS:
Overall Officials: Gail Darling, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No